CLINICAL TRIAL: NCT03457714
Title: Guided Internet Delivered Cognitive-Behaviour Therapy for Persons With Spinal Cord Injury: A Feasibility Trial
Status: Completed | Type: Observational
Sponsor: University of Regina (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-104
Record Dates: First submitted 2017-12-07; First posted 2018-03-07 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Spinal Cord Injuries; Depression; Anxiety
Keywords: spinal cord injuries; anxiety; depression; internet-delivered cognitive behaviour therapy; pilot study
MeSH Terms: conditions — Spinal Cord Injuries; Depression; Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Guided I-CBT for persons with SCI: Persons with spinal cord injury
  Interventions: Behavioral: Guided ICBT for persons with Spinal Cord Injury; Other: Survey

INTERVENTIONS:
Behavioral: Guided ICBT for persons with Spinal Cord Injury — An 8-week guided internet-delivered cognitive behavioural therapy (ICBT) will be delivered to participants who have sustained a spinal cord injury. In addition to the online program, a guide with experience delivering ICBT will provide support by email or telephone once a week. The guide will spend approximately 15 minutes per week/per client.
Other: Survey — Caregiver burden and mental health will be assessed through online questionnaires.

SUMMARY:
In Canada the prevalence of spinal cord injury (SCI) is approximately 85,556, with incidence rates of traumatic and non-traumatic SCI at 1,785 and 2,286 cases per year, respectively. Common secondary health conditions experienced by individuals with SCI include psychological distress and pain. Appropriate management of these secondary conditions, through a multidisciplinary approach, is imperative as they have been shown to contribute to slower recovery, increased negative outcomes, and greater rates of rehospitalizations and health care utilization. However, resource limitations can restrict the ability of service providers to deliver these integrative biopsychosocial approaches in the community. In Canada over 37% of individuals with SCI expressed a need for emotional counselling; of these, only 43% felt that these needs were met. Transportation can also be a significant issue for persons with SCI, with 87% and 73% respectively expressing a need for short- and long-distance transportation. Guided internet delivered cognitive behavioural therapy (ICBT) program offers an alternative approach for psychosocial service delivery in the community. The program provides online structured self-help modules based on the principles of cognitive behavioural therapy (CBT) in combination with guidance from a coach through weekly emails and telephone calls. ICBT has shown to have a greater reduction in levels of anxiety and depression post treatment compared to a waitlist control group, and these levels were maintained at both 3 and 12 month follow-ups. ICBT was shown to have similar effects to face-to-face CBT. These studies demonstrate that guided ICBT is a safe and effective alternative to face-to-face interventions and it may be beneficial for under serviced populations. Hence, examination of its effectiveness is warranted in the SCI population which faces various psychological and somatic secondary issues. Participants with SCI will receive a 8 week guided ICBT program called the Chronic Conditions Course for persons with SCI. The program is completed over 8 weeks with once a week guidance from a coach. The guided course consists of five lessons, "Do It Yourself" activities, and case vignettes adapted from persons with SCI. The course also provides guidance and resources on other essential skills for persons with SCI, including communicating with health care professional, managing chronic pain, and sleep hygiene. Psychosocial outcomes will be assessed at baseline, 8 weeks, and at 3 months. Data on intervention usage and satisfaction measures will also be examined through a qualitative interview. Caregivers of participants will be asked to complete self-report measures and a qualitative interview regarding their caregiver burden.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* residing in Canada
* diagnosed with spinal cord injury
* able to access a computer and internet service
* willing to provide a physician as emergency contact

Exclusion Criteria:

* high suicide risk
* suicide attempt or hospitalization in the last year
* primary problems with psychosis, alcohol or drug problems, mania
* currently receiving active psychological treatment for anxiety or depression
* not present in Canada during treatment
* concerns about online therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any individual with a spinal cord injury will be recruited through primary care physicians, rehabilitation facilities, and community peer groups.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Change in depression | baseline, start of each Lesson 2-5, 8 weeks, 3 months
  Patient Health Questionnaire - 9 Item (PHQ-9). Higher total scores indicate greater severity of depression. Scores range from 0 to 27.
Change in anxiety | baseline, start of each Lesson 2-5, 8 weeks, 3 months
  Generalize Anxiety Disorder - 7 Item (GAD7). Higher total scores indicate greater severity of anxiety. Scores range from 0 to 21
Change in Caregiver Burden from baseline to 8 weeks (Caregivers of persons with SCI only) | baseline, 8 weeks
  Caregiver burden questionnaire. The tool has 12 items. Total scores ranging from 0 to 18. Higher scores indicate greater burden

SECONDARY OUTCOMES:
Pain (Persons with SCI only) | baseline, 8 weeks, 3 months
  International Spinal Cord Injury Pain Basic Data Set v2.0 ISCIPBDS
Pain interference (Persons with SCI only) | baseline, 8 weeks, 3 months
  Brief Pain Inventory Short Form; BPI-SF
Quality of life (Persons with SCI only) | baseline, 8 weeks, 3 months
  Spinal Cord Injury Quality of Life Short Form; SCI-QoL-SF
Service usage (Persons with SCI only) | baseline, 8 weeks, 3 months
Quality of Life (Caregivers of persons with SCI only) | baseline, 8 weeks, 3 months, 6 months, and 1 year follow up
  EQ5D

CONTACTS AND LOCATIONS:
Overall Officials: Swati Mehta, PhD, Principal Investigator — University of Regina; Heather D Hadjistavropoulos, PhD, Study Director — University of Regina
Locations (1):
- Online Therapy Unit, University of Regina, Regina, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mehta S, Hadjistavropoulos HD, Earis D, Titov N, Dear BF. Patient perspectives of Internet-delivered cognitive behavior therapy for psychosocial issues post spinal cord injury. Rehabil Psychol. 2019 Aug;64(3):351-359. doi: 10.1037/rep0000276. Epub 2019 Apr 8. PMID 30958020